CLINICAL TRIAL: NCT06297343
Title: Study of the Risk of Ischaemia Following the Creation of an Arteriovenous Fistula
Acronym: MODIFVASC
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A02491-44
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with chronic renal failure: Adult patients with chronic renal failure for whom arteriovenous fistula creation is planned
  Interventions: Procedure: Creation of an arteriovenous fistula

INTERVENTIONS:
Procedure: Creation of an arteriovenous fistula — Patients will undergo the surgical procedure to create an arteriovenous fistula and will be discharged the same day (outpatient care, or an overnight stay in hospital if they live a long way from the hospital, have multiple pathologies or are socially isolated). An arteriovenous fistula is created under local or general anaesthetic. On the day of the operation, the type of arteriovenous fistula created, the side of the arteriovenous fistula, the location of the arteriovenous fistula and the patency of the arteriovenous fistula will be collected.

SUMMARY:
The purpose of this study is to identify functional vascular changes and clinical factors correlated with the occurrence of short- or medium-term hand ischaemia after arteriovenous fistula creation.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, non-randomised, descriptive, single-centre study with no comparator.

The study population will be adult patients with chronic renal failure for whom an arteriovenous fistula has been planned.

Patients requiring the creation of an arteriovenous fistula by the surgeons at Hôpital Privé des Peupliers will be seen beforehand in the usual pre-operative consultation, during which the surgeon will explain the principle of the operation and the expected benefits/risks. On the day of surgery, patients will undergo the surgical procedure to create an arteriovenous fistula and will be discharged the same day. Patients will be reviewed during post-operative follow-up visits at 1, 6 and 12 months as in standard practice. All the data collected in the study were collected in routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Stage 5 chronic kidney disease, on dialysis or not on dialysis;
* Requiring the creation of an arteriovenous fistula;
* Membership of a social insurance scheme;
* Patient having been informed and having formulated his/her oral non-opposition to participate in the research.

Exclusion Criteria:

* Contraindication to the proposed surgery ;
* Reduced life expectancy in the opinion of the investigator;
* Medical or biological conditions which, in the opinion of the investigator, could influence the interpretation of the results of the study or the safety of the patient;
* Patient uncooperative with protocol requirements or unable to attend scheduled visits to the centre;
* Other surgical or medical intervention planned during the study;
* Pregnant or likely to be pregnant (of childbearing age, without effective contraception) or breastfeeding;
* Participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient under guardianship or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult patients suffering from chronic renal failure for whom the creation of an arteriovenous fistula is planned.
Sampling Method: Non-Probability Sample
Enrollment: 544 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of ischaemia of the hand | 12 months
  Number and proportion of patients with ischaemia (Yes = stages 1, 2 or 3/No = stage 0) according to the preoperative American Vascular Surgery ischaemia classification :
  0 - nothing
  1. - cold hand
  2. - pain on exercise and/or during dialysis
  3. - permanent pain, wound (ulceration, necrosis, gangrene)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé des Peupliers, Paris, France